CLINICAL TRIAL: NCT00793624
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of 48 Weeks of Once Daily Treatment of Orally Inhaled BI 1744 CL (5 µg [2 Actuations of 2.5 ug] and 10 ug [2 Actuations of 5 ug]) Delivered by the Respimat® Inhaler, and 48 Weeks of Twice Daily Foradil® (12 µg) Delivered by the Aerolizer® Inhaler, in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Safety and Efficacy of BI 1744 CL in Patients With Chronic Obstructive Pulmonary Disease I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.13; 2008-001933-84 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Formoterol Fumarate

ARMS (4):
- Olodaterol (BI 1744) Low (Experimental): Low dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744)
- Olodaterol (BI 1744) High (Experimental): High dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744)
- Formoterol 12mcg (Active Comparator): 12mcg inhaled twice daily from the Aerolizer inhaler
  Interventions: Drug: Formoterol
- Placebo (Placebo Comparator): Olodaterol (BI 1744) placebo inhaled once daily from the Respimat inhaler and/or Formoterol placebo inhaled twice daily from the Aerolizer inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olodaterol (BI 1744) — Comparison of low and high doses on efficacy and safety in COPD patients
  Arms: Olodaterol (BI 1744) Low
Drug: Olodaterol (BI 1744) — Comparison of low and high doses on efficacy and safety in COPD patients
  Arms: Olodaterol (BI 1744) High
Drug: Formoterol — Active comparator with Olodaterol (BI 1744) on safety and efficacy in COPD patients
  Arms: Formoterol 12mcg
Drug: Placebo — Placebo for comparison with Olodaterol (BI 1744) on safety and efficacy in COPD patients
  Arms: Placebo
Drug: Placebo — Placebo for comparison Formoterolon safety and efficacy in COPD patients
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the long-term efficacy and safety of once daily treatment of BI 1744 CL inhalation solution (5 and 10 mcg) delivered via the Respimat® inhaler, in patients with COPD.

ELIGIBILITY:
Inclusion criteria:

1. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:post-bronchodilator FEV1<80% of predicted normal (ECSC) and a post-bronchodilator FEV1/FVC <70% at Visit 1
2. Male or female patients, 40 years of age or older
3. Patients must be current or ex-smokers with a smoking history of more than 10 pack years:

Exclusion criteria:

1. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an SGOT >x2 ULN, SGPT >x2 ULN, bilirubin >x2 ULN or creatinine >x2 ULN
2. Patients with a history of asthma and/or total blood eosinophil count greater than 600/mm3
3. Patients with thyrotoxicosis, paroxysmal tachycardia (>100 beats per minute)
4. Patients with a history of myocardial infarction within 1 year of screening visit, unstable or life-threatening cardiac arrhythmia, hospitalization for heart failure within the past year, known active tuberculosis, a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years, life-threatening pulmonary obstruction, cystic fibrosis, clinically evident bronchiectasis, significant alcohol or drug abuse
5. Patients who have undergone thoracotomy with pulmonary resection
6. Patients being treated with oral beta-adrenergics or oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
7. Patients who regularly use daytime oxygen therapy for more than one hour per day.
8. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program
9. Pregnant or nursing women
10. Women of childbearing potential not using two effective methods of birth control (one barrier and one non-barrier).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 906 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (93):
- Argentina (4):
  - 1222.13.2401 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1222.13.2403 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1222.13.2402 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1222.13.2404 Boehringer Ingelheim Investigational Site, Monte Grande
- Brazil (5):
  - 1222.13.2502 Boehringer Ingelheim Investigational Site, Juiz de Fora
  - 1222.13.2503 Boehringer Ingelheim Investigational Site, Rio de Janeiro
  - 1222.13.2505 Boehringer Ingelheim Investigational Site, Rio de Janeiro
  - 1222.13.2501 Boehringer Ingelheim Investigational Site, São Paulo
  - 1222.13.2504 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (11):
  - 1222.13.1408 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1222.13.1407 Boehringer Ingelheim Investigational Site, Chilliwack, British Columbia
  - 1222.13.1403 Boehringer Ingelheim Investigational Site, Downsview, Ontario
  - 1222.13.1412 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1222.13.1401 Boehringer Ingelheim Investigational Site, Niagara Falls, Ontario
  - 1222.13.1410 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1222.13.1413 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1222.13.1404 Boehringer Ingelheim Investigational Site, La Malbaie, Quebec
  - 1222.13.1411 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1222.13.1406 Boehringer Ingelheim Investigational Site, Point Claire, Quebec
  - 1222.13.1402 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Croatia (4):
  - 1222.13.3502 Boehringer Ingelheim Investigational Site, Dubrovnik
  - 1222.13.3503 Boehringer Ingelheim Investigational Site, Rijeka
  - 1222.13.3504 Boehringer Ingelheim Investigational Site, Split
  - 1222.13.3501 Boehringer Ingelheim Investigational Site, Zagreb
- Czechia (3):
  - 1222.13.3401 Boehringer Ingelheim Investigational Site, Beroun
  - 1222.13.3403 Boehringer Ingelheim Investigational Site, Český Těšín
  - 1222.13.3402 Boehringer Ingelheim Investigational Site, Tábor
- Denmark (3):
  - 1222.13.2003 Boehringer Ingelheim Investigational Site, Aalborg
  - 1222.13.2002 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1222.13.2001 Boehringer Ingelheim Investigational Site, Silkeborg
- Finland (3):
  - 1222.13.2103 Boehringer Ingelheim Investigational Site, Lahti
  - 1222.13.2101 Boehringer Ingelheim Investigational Site, Tampere
  - 1222.13.2102 Boehringer Ingelheim Investigational Site, Turku
- Germany (12):
  - 1222.13.1502 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.13.1503 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.13.1506 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.13.1501 Boehringer Ingelheim Investigational Site, Cologne
  - 1222.13.1511 Boehringer Ingelheim Investigational Site, Dortmund
  - 1222.13.1514 Boehringer Ingelheim Investigational Site, Essen
  - 1222.13.1509 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1222.13.1508 Boehringer Ingelheim Investigational Site, Hanover
  - 1222.13.1510 Boehringer Ingelheim Investigational Site, Hanover
  - 1222.13.1512 Boehringer Ingelheim Investigational Site, Kiel
  - 1222.13.1505 Boehringer Ingelheim Investigational Site, Reinfeld
  - 1222.13.1507 Boehringer Ingelheim Investigational Site, Schwerin
- 1222.13.2901 Boehringer Ingelheim Investigational Site, Kowloon, Hong Kong
- India (11):
  - 1222.13.2804 Boehringer Ingelheim Investigational Site, Bangalore
  - 1222.13.2803 Boehringer Ingelheim Investigational Site, Chennai
  - 1222.13.2806 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1222.13.2810 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1222.13.2801 Boehringer Ingelheim Investigational Site, Indore
  - 1222.13.2807 Boehringer Ingelheim Investigational Site, Indore
  - 1222.13.2805 Boehringer Ingelheim Investigational Site, Jaipur
  - 1222.13.2802 Boehringer Ingelheim Investigational Site, Ludhiana, Punjab
  - 1222.13.2809 Boehringer Ingelheim Investigational Site, Mumbai
  - 1222.13.2812 Boehringer Ingelheim Investigational Site, Mumbai
  - 1222.13.2811 Boehringer Ingelheim Investigational Site, Pune
- Italy (5):
  - 1222.13.1704 Boehringer Ingelheim Investigational Site, Catania
  - 1222.13.1702 Boehringer Ingelheim Investigational Site, Genova
  - 1222.13.1701 Boehringer Ingelheim Investigational Site, Pisa
  - 1222.13.1705 Boehringer Ingelheim Investigational Site, Siena
  - 1222.13.1703 Boehringer Ingelheim Investigational Site, Trieste
- Malaysia (4):
  - 1222.13.3103 Boehringer Ingelheim Investigational Site, Batu Caves
  - 1222.13.3101 Boehringer Ingelheim Investigational Site, Kota Kinabalu
  - 1222.13.3102 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1222.13.3104 Boehringer Ingelheim Investigational Site, Kuantan
- Norway (2):
  - 1222.13.2201 Boehringer Ingelheim Investigational Site, Bergen
  - 1222.13.2202 Boehringer Ingelheim Investigational Site, Oslo
- Philippines (3):
  - 1222.13.3203 Boehringer Ingelheim Investigational Site, Cebu
  - 1222.13.3201 Boehringer Ingelheim Investigational Site, Quezon City
  - 1222.13.3202 Boehringer Ingelheim Investigational Site, Quezon City
- South Africa (2):
  - 1222.13.2302 Boehringer Ingelheim Investigational Site, Durban
  - 1222.13.2301 Boehringer Ingelheim Investigational Site, Pretoria
- South Korea (6):
  - 1222.13.2701 Boehringer Ingelheim Investigational Site, Gwangju
  - 1222.13.2702 Boehringer Ingelheim Investigational Site, Incheon
  - 1222.13.2703 Boehringer Ingelheim Investigational Site, Seoul
  - 1222.13.2705 Boehringer Ingelheim Investigational Site, Seoul
  - 1222.13.2706 Boehringer Ingelheim Investigational Site, Seoul
  - 1222.13.2704 Boehringer Ingelheim Investigational Site, Suwon
- Spain (6):
  - 1222.13.1803 Boehringer Ingelheim Investigational Site, Aranjuez
  - 1222.13.1806 Boehringer Ingelheim Investigational Site, Elda
  - 1222.13.1802 Boehringer Ingelheim Investigational Site, els Hostalets de Balenyà
  - 1222.13.1804 Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón
  - 1222.13.1805 Boehringer Ingelheim Investigational Site, Valladolid
  - 1222.13.1801 Boehringer Ingelheim Investigational Site, Vic (Barcelona)
- Sweden (2):
  - 1222.13.1901 Boehringer Ingelheim Investigational Site, Boden
  - 1222.13.1902 Boehringer Ingelheim Investigational Site, Sundsvall
- Thailand (3):
  - 1222.13.3302 Boehringer Ingelheim Investigational Site, Bangkok
  - 1222.13.3303 Boehringer Ingelheim Investigational Site, Bangkok
  - 1222.13.3301 Boehringer Ingelheim Investigational Site, Chiang Mai
- Ukraine (3):
  - 1222.13.3602 Boehringer Ingelheim Investigational Site, Ivano-Frankivsk
  - 1222.13.3601 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1222.13.3603 Boehringer Ingelheim Investigational Site, Kiev

REFERENCES:
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Andreas S, Bothner U, de la Hoz A, Kloer I, Trampisch M, Alter P. A Post Hoc Holter ECG Analysis of Olodaterol and Formoterol in Moderate-to-Very-Severe COPD. Int J Chron Obstruct Pulmon Dis. 2020 Aug 10;15:1955-1965. doi: 10.2147/COPD.S246353. eCollection 2020. PMID 32848381
- [Derived] Andreas S, Bothner U, Trampisch M, Haensel M, Buhl R, Alter P. Effect of long-acting beta2-agonists olodaterol and formoterol on heart rate and blood pressure in chronic obstructive pulmonary disease patients. Pulm Pharmacol Ther. 2018 Oct;52:1-6. doi: 10.1016/j.pupt.2018.08.002. Epub 2018 Aug 2. PMID 30077810
- [Derived] Koch A, Pizzichini E, Hamilton A, Hart L, Korducki L, De Salvo MC, Paggiaro P. Lung function efficacy and symptomatic benefit of olodaterol once daily delivered via Respimat(R) versus placebo and formoterol twice daily in patients with GOLD 2-4 COPD: results from two replicate 48-week studies. Int J Chron Obstruct Pulmon Dis. 2014 Jul 5;9:697-714. doi: 10.2147/COPD.S62502. eCollection 2014. PMID 25045258

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were randomized but not treated due to withdrawn consent and inability to perform spirometry prior to dosing.
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler.
- Olodaterol (Olo) 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olodaterol (Olo) 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Form 12 mcg: Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler.
Period: Overall Study
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd | Form 12 mcg
Started | 225 | 227 | 225 | 227
Completed | 168 | 191 | 186 | 184
Not Completed | 57 | 36 | 39 | 43
Not completed — Adverse Event | 18 | 16 | 15 | 20
Not completed — Lost to Follow-up | 2 | 2 | 4 | 0
Not completed — Withdrawal by Subject | 20 | 9 | 11 | 14
Not completed — Lack of Efficacy | 9 | 2 | 1 | 3
Not completed — Non compliance with protocol | 2 | 3 | 2 | 3
Not completed — Other reason not described above | 6 | 4 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Total: Total of all reporting groups
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg | Total
Number analyzed (Participants) | 225 | 227 | 225 | 227 | 904
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.4) | 63.7 (9.1) | 62.6 (8.8) | 64.8 (8.6) | 63.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 50 | 55 | 48 | 198
  Male | 180 | 177 | 170 | 179 | 706
Tiotropium (Tio) Use Stratum [Number; unit: Number of participants]
  Non-tiotropium | 169 | 168 | 167 | 169 | 673
  Tiotropium | 56 | 59 | 58 | 58 | 231

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 24 Weeks
Description: Response was defined as change from baseline. Baseline FEV1 was defined as the mean of the -1 h and -10 min measurements performed just prior to administration of the first am dose of randomized treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit interaction as fixed categorical effects, baseline and baseline-by-visit interaction as fixed continuous covariates and patient as random effect. FEV1 AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Week 24
Population: Full analysis set (FAS). FAS is defined as all randomized patients who received at least one dose of treatment and had both baseline data and at least one post-baseline measurement at or before 24 weeks for any of the co-primary efficacy variables.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | -0.009 (0.016) | 0.142 (0.015) | 0.156 (0.015) | 0.168 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects,baseline, baseline-by-visit as fixed covariates, patient as random effect; Mean Difference (Final Values) = 0.151, 95% CI [0.110 to 0.193], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.165, 95% CI [0.124 to 0.206], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.177, 95% CI [0.136 to 0.218], Standard Error of Mean 0.021 — Form 12 mcg minus Placebo

2. Primary Outcome: Trough FEV1 Response at Week 24
Description: Response was defined as change from baseline. Baseline trough FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FEV1 is defined as the FEV1 performed at -10 mins prior to study drug inhalation as the end of the dosing interval or the mean of -1h and -10 min FEV1s if both available. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 24.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.056 (0.015) | 0.021 (0.015) | 0.028 (0.015) | -0.002 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.078, 95% CI [0.037 to 0.118], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.085, 95% CI [0.044 to 0.125], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0088, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.054, 95% CI [0.014 to 0.095], Standard Error of Mean 0.021 — Form 12 mcg minus Placebo

3. Primary Outcome: Mahler Transitional Dyspnea Index Focal Score at 24 Weeks
Description: Mahler Transitional Dyspnea Index (TDI) focal score measures 3 components of dyspnea that evoke dyspnea in daily living: Functional Impairment, Magnitude of Task, and Magnitude of Effort. The TDI measures the change from the baseline assessment ranging from -9 (most deterioration) to +9 (most improvement).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 192 | 212 | 207 | 202
score on a scale | 2.046 (0.255) | 2.234 (0.240) | 2.068 (0.245) | 1.818 (0.247)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.5843, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.188, 95% CI [-0.485 to 0.860], Standard Error of Mean 0.343 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.9494, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.022, 95% CI [-0.656 to 0.699], Standard Error of Mean 0.345 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.5099, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.288, 95% CI [-0.908 to 0.451], Standard Error of Mean 0.346 — Form 12 mcg minus Placebo

4. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score at 24 Weeks
Description: Saint George's Respiratory Questionnaire (SGRQ) measures the impact of COPD on overall health, daily life, and perceived well-being ranging from 0 (no limitations) to 100 (most limitations).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 185 | 200 | 202 | 202
score on a scale | 41.068 (1.038) | 38.627 (0.995) | 37.674 (0.998) | 40.116 (0.994)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0816, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.442, 95% CI [-5.190 to 0.307], Standard Error of Mean 1.401 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0155, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.394, 95% CI [-6.141 to -0.648], Standard Error of Mean 1.400 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.4954, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.952, 95% CI [-3.691 to 1.787], Standard Error of Mean 1.396 — Form 12 mcg minus Placebo

5. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score at 12 Weeks
Description: as for outcome 4
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 185 | 200 | 202 | 202
score on a scale | 42.105 (1.027) | 39.320 (0.986) | 36.961 (0.989) | 40.351 (0.992)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0450, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.785, 95% CI [-5.507 to -0.063], Standard Error of Mean 1.387 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.144, 95% CI [-7.864 to -2.425], Standard Error of Mean 1.386 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.2061, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.754, 95% CI [-4.474 to 0.966], Standard Error of Mean 1.386 — Form 12 mcg minus Placebo

6. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score at 48 Weeks
Description: as for outcome 4
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 185 | 200 | 202 | 202
score on a scale | 40.415 (1.057) | 38.545 (1.000) | 36.850 (1.015) | 40.431 (1.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1878, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.871, 95% CI [-4.655 to 0.914], Standard Error of Mean 1.419 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0126, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.565, 95% CI [-6.364 to -0.767], Standard Error of Mean 1.427 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.9913, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.016, 95% CI [-2.782 to 2.814], Standard Error of Mean 1.426 — Form 12 mcg minus Placebo

7. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score at 24 Weeks for Combined Analysis
Description: Saint George's Respiratory Questionnaire (SGRQ) measures the impact of COPD on overall health, daily life, and perceived well-being ranging from 0 (no limitations) to 100 (most limitations). This is a combined analysis of the data from NCT00793624 and NCT00796653 showing adjusted values using a MMRM model.
Time Frame: Baseline, Week 24
Population: Full analysis sets (FAS) of the trials NCT00793624 and NCT00796653. FAS is defined as all randomized patients who received at least one dose of treatment and had both baseline data and at least one post-baseline measurement at or before 24 weeks for any of the co-primary efficacy variables.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 387 | 416 | 414 | 408
score on a scale | 41.639 (0.718) | 38.794 (0.693) | 38.205 (0.695) | 40.391 (0.699)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Olo 5 mcg qd minus Placebo; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis; Mean Difference (Final Values) = -2.846, 95% CI [-4.751 to -0.940], Standard Error of Mean 0.972 — Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects,baseline, baseline-by-visit as fixed covariates, patient as random effect
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Olo 10 mcg qd minus Placebo; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = -3.434, 95% CI [-5.343 to -1.525], Standard Error of Mean 0.973 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Form 10 mcg qd minus Placebo; Test type: Superiority or Other; p = 0.2009, Mixed Models Analysis; Mean Difference (Final Values) = -1.248, 95% CI [-3.161 to 0.665], Standard Error of Mean 0.976 — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 2 Weeks
Description: as for outcome 1
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.015 (0.015) | 0.201 (0.015) | 0.181 (0.015) | 0.221 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.186, 95% CI [0.146 to 0.226], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.166, 95% CI [0.126 to 0.206], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.206, 95% CI [0.166 to 0.246], Standard Error of Mean 0.020 — Form 12 mcg minus Placebo

9. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 6 Weeks
Description: as for outcome 1
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.001 (0.015) | 0.178 (0.015) | 0.161 (0.015) | 0.194 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.176, 95% CI [0.136 to 0.217], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.160, 95% CI [0.119 to 0.200], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.192, 95% CI [0.152 to 0.233], Standard Error of Mean 0.021 — Form 12 mcg minus Placebo

10. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 12 Weeks
Description: as for outcome 1
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | -0.003 (0.015) | 0.176 (0.015) | 0.167 (0.015) | 0.182 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.178, 95% CI [0.137 to 0.219], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.170, 95% CI [0.129 to 0.211], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.185, 95% CI [0.144 to 0.226], Standard Error of Mean 0.021 — Form 12 mcg minus Placebo

11. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 48 Weeks
Description: as for outcome 1
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | -0.023 (0.016) | 0.122 (0.015) | 0.123 (0.015) | 0.149 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.145, 95% CI [0.103 to 0.186], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.146, 95% CI [0.105 to 0.188], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.172, 95% CI [0.130 to 0.214], Standard Error of Mean 0.021 — Form 12 mcg minus Placebo

12. Secondary Outcome: Trough FEV1 Response at Week 2
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 2.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.019 (0.015) | 0.068 (0.014) | 0.060 (0.014) | 0.061 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.087, 95% CI [0.048 to 0.126], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.079, 95% CI [0.040 to 0.118], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.080, 95% CI [0.040 to 0.119], Standard Error of Mean 0.020 — Form 12 mcg minus Placebo

13. Secondary Outcome: Trough FEV1 Response at Week 6
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 6.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.037 (0.015) | 0.049 (0.014) | 0.041 (0.014) | 0.042 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.086, 95% CI [0.047 to 0.125], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.078, 95% CI [0.038 to 0.117], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.079, 95% CI [0.039 to 0.119], Standard Error of Mean 0.020 — Form 12 mcg minus Placebo

14. Secondary Outcome: Trough FEV1 Response at Week 12
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 12.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.027 (0.015) | 0.056 (0.014) | 0.048 (0.014) | 0.033 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.083, 95% CI [0.043 to 0.123], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.075, 95% CI [0.035 to 0.114], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0037, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.059, 95% CI [0.019 to 0.100], Standard Error of Mean 0.020 — Form 12 mcg minus Placebo

15. Secondary Outcome: Trough FEV1 Response at Week 18
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 18.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.019 (0.015) | 0.046 (0.014) | 0.026 (0.015) | 0.023 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.065, 95% CI [0.025 to 0.105], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0276, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.045, 95% CI [0.005 to 0.085], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0426, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.042, 95% CI [0.001 to 0.082], Standard Error of Mean 0.021 — Form 12 mcg minus Placebo

16. Secondary Outcome: Trough FEV1 Response at Week 32
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 32.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.023 (0.015) | 0.023 (0.015) | 0.026 (0.015) | 0.021 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0237, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.047, 95% CI [0.006 to 0.087], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0175, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.049, 95% CI [0.009 to 0.090], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0339, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.044, 95% CI [0.003 to 0.085], Standard Error of Mean 0.021 — Form 12 mcg minus Placebo

17. Secondary Outcome: Trough FEV1 Response at Week 40
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 40.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.020 (0.016) | 0.020 (0.015) | 0.017 (0.015) | 0.004 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0537, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.040, 95% CI [-0.001 to 0.081], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0808, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.037, 95% CI [-0.004 to 0.078], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.2579, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.024, 95% CI [-0.017 to 0.065], Standard Error of Mean 0.021 — Form 12 mcg minus Placebo

18. Secondary Outcome: Trough FEV1 Response at Week 48
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug at week 48.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.065 (0.015) | 0.003 (0.015) | -0.009 (0.015) | -0.006 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.068, 95% CI [0.027 to 0.109], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0069, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.059, 95% CI [0.018 to 0.101], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.080, 95% CI [0.040 to 0.119], Standard Error of Mean 0.020 — Form 12 mcg minus Placebo

19. Secondary Outcome: Peak FEV1 (0-3h) Response After 2 Weeks
Description: Response was defined as change from baseline. Baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values prior to first dose of randomized treatment. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.100 (0.016) | 0.277 (0.016) | 0.250 (0.016) | 0.290 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.177, 95% CI [0.135 to 0.220], Standard Error of Mean 0.022 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.150, 95% CI [0.108 to 0.193], Standard Error of Mean 0.022 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.190, 95% CI [0.148 to 0.233], Standard Error of Mean 0.022 — Form 12 mcg minus Placebo

20. Secondary Outcome: Peak FEV1 (0-3h) Response After 6 Weeks
Description: as for outcome 19
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.081 (0.016) | 0.248 (0.016) | 0.234 (0.016) | 0.264 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.166, 95% CI [0.124 to 0.209], Standard Error of Mean 0.022 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.152, 95% CI [0.109 to 0.195], Standard Error of Mean 0.022 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.182, 95% CI [0.139 to 0.226], Standard Error of Mean 0.022 — Form 12 mcg minus Placebo

21. Secondary Outcome: Peak FEV1 (0-3h) Response After 12 Weeks
Description: as for outcome 19
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.082 (0.016) | 0.247 (0.016) | 0.241 (0.016) | 0.256 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.165, 95% CI [0.122 to 0.208], Standard Error of Mean 0.022 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.159, 95% CI [0.116 to 0.203], Standard Error of Mean 0.022 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.174, 95% CI [0.130 to 0.218], Standard Error of Mean 0.022 — Form 12 mcg minus Placebo

22. Secondary Outcome: Peak FEV1 (0-3h) Response After 24 Weeks
Description: as for outcome 19
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.068 (0.017) | 0.216 (0.016) | 0.225 (0.016) | 0.236 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.148, 95% CI [0.104 to 0.191], Standard Error of Mean 0.022 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.167, 95% CI [0.112 to 0.200], Standard Error of Mean 0.022 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.167, 95% CI [0.123 to 0.211], Standard Error of Mean 0.022 — Form 12 mcg minus Placebo

23. Secondary Outcome: Peak FEV1 (0-3h) Response After 48 Weeks
Description: as for outcome 19
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 48 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.053 (0.017) | 0.192 (0.016) | 0.193 (0.016) | 0.215 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.139, 95% CI [0.095 to 0.183], Standard Error of Mean 0.023 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.140, 95% CI [0.095 to 0.184], Standard Error of Mean 0.023 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.162, 95% CI [0.117 to 0.206], Standard Error of Mean 0.023 — Form 12 mcg minus Placebo

24. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 2 Weeks
Description: Response was defined as change from baseline. Baseline FVC was defined as the mean of the -1 h and -10 min measurements performed just prior to administration of the first am dose of randomized treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit interaction as fixed categorical effects, baseline and baseline-by-visit interaction as fixed continuous covariates and patient as random effect. FVC AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.076 (0.028) | 0.299 (0.027) | 0.311 (0.027) | 0.383 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.223, 95% CI [0.149 to 0.297], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.235, 95% CI [0.161 to 0.309], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.307, 95% CI [0.233 to 0.381], Standard Error of Mean 0.038 — Form 12 mcg minus Placebo

25. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 6 Weeks
Description: as for outcome 24
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.016 (0.028) | 0.252 (0.027) | 0.265 (0.027) | 0.326 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.236, 95% CI [0.161 to 0.310], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.249, 95% CI [0.175 to 0.324], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.310, 95% CI [0.235 to 0.384], Standard Error of Mean 0.038 — Form 12 mcg minus Placebo

26. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 12 Weeks
Description: as for outcome 24
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.023 (0.028) | 0.233 (0.027) | 0.278 (0.027) | 0.300 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.210, 95% CI [0.135 to 0.285], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.254, 95% CI [0.179 to 0.329], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.276, 95% CI [0.201 to 0.352], Standard Error of Mean 0.039 — Form 12 mcg minus Placebo

27. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 24 Weeks
Description: as for outcome 24
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.037 (0.029) | 0.220 (0.027) | 0.252 (0.028) | 0.279 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.182, 95% CI [0.107 to 0.258], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.215, 95% CI [0.139 to 0.291], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.242, 95% CI [0.166 to 0.318], Standard Error of Mean 0.039 — Form 12 mcg minus Placebo

28. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at 48 Weeks
Description: as for outcome 24
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.016 (0.029) | 0.196 (0.028) | 0.219 (0.028) | 0.260 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.179, 95% CI [0.103 to 0.256], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.203, 95% CI [0.126 to 0.280], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.243, 95% CI [0.166 to 0.320], Standard Error of Mean 0.039 — Form 12 mcg minus Placebo

29. Secondary Outcome: Trough FVC Response at Week 2
Description: Response was defined as change from baseline. Baseline trough FVC was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FVC is defined as the FVC performed at -10 mins prior to study drug inhalation as the end of the dosing interval or the mean of -1h and -10 min FVCs if both available. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | 0.042 (0.028) | 0.110 (0.027) | 0.119 (0.028) | 0.126 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0781, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.068, 95% CI [-0.008 to 0.143], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0455, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.077, 95% CI [0.002 to 0.153], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0290, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.085, 95% CI [0.009 to 0.160], Standard Error of Mean 0.039 — Form 12 mcg minus Placebo

30. Secondary Outcome: Trough FVC Response at Week 6
Description: as for outcome 29
Time Frame: as for outcome 13
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.046 (0.029) | 0.065 (0.027) | 0.085 (0.028) | 0.090 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0043, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.110, 95% CI [0.035 to 0.186], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.131, 95% CI [0.055 to 0.207], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.136, 95% CI [0.060 to 0.212], Standard Error of Mean 0.039 — Form 12 mcg minus Placebo

31. Secondary Outcome: Trough FVC Response at Week 12
Description: as for outcome 29
Time Frame: as for outcome 14
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.018 (0.029) | 0.079 (0.028) | 0.087 (0.028) | 0.068 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0136, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.097, 95% CI [0.020 to 0.173], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0076, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.105, 95% CI [0.028 to 0.182], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0294, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.086, 95% CI [0.009 to 0.163], Standard Error of Mean 0.039 — Form 12 mcg minus Placebo

32. Secondary Outcome: Trough FVC Response at Week 18
Description: as for outcome 29
Time Frame: as for outcome 15
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | 0.060 (0.029) | 0.066 (0.028) | 0.078 (0.028) | 0.063 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.8674, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.007, 95% CI [-0.071 to 0.084], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6487, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.018, 95% CI [-0.060 to 0.096], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.9267, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.004, 95% CI [-0.074 to 0.081], Standard Error of Mean 0.040 — Form 12 mcg minus Placebo

33. Secondary Outcome: Trough FVC Response at Week 24
Description: as for outcome 29
Time Frame: as for outcome 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.018 (0.029) | 0.038 (0.028) | 0.064 (0.028) | 0.001 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1603, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.056, 95% CI [-0.022 to 0.134], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0399, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.082, 95% CI [0.004 to 0.160], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.6328, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.019, 95% CI [-0.059 to 0.098], Standard Error of Mean 0.040 — Form 12 mcg minus Placebo

34. Secondary Outcome: Trough FVC Response at Week 32
Description: as for outcome 29
Time Frame: as for outcome 16
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | 0.019 (0.030) | 0.080 (0.028) | 0.084 (0.028) | 0.077 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1270, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.061, 95% CI [-0.017 to 0.139], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1076, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.064, 95% CI [-0.014 to 0.143], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.1492, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.058, 95% CI [-0.021 to 0.137], Standard Error of Mean 0.040 — Form 12 mcg minus Placebo

35. Secondary Outcome: Trough FVC Response at Week 48
Description: as for outcome 29
Time Frame: as for outcome 18
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | -0.061 (0.030) | 0.022 (0.028) | -0.002 (0.029) | 0.006 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0385, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.083, 95% CI [0.004 to 0.162], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1420, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.059, 95% CI [-0.020 to 0.138], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0965, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.067, 95% CI [-0.012 to 0.147], Standard Error of Mean 0.040 — Form 12 mcg minus Placebo

36. Secondary Outcome: Trough FVC Response at Week 40
Description: as for outcome 29
Time Frame: as for outcome 17
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 205 | 220 | 219 | 215
Liter | 0.028 (0.030) | 0.087 (0.028) | 0.086 (0.028) | 0.052 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1394, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.059, 95% CI [-0.019 to 0.138], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1532, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.058, 95% CI [-0.022 to 0.137], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.5511, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.024, 95% CI [-0.055 to 0.104], Standard Error of Mean 0.041 — Form 12 mcg minus Placebo

37. Secondary Outcome: Peak FVC (0-3h) Response After 2 Weeks
Description: Response was defined as change from baseline. Baseline peak FVC was defined as the mean of the available pre-dose peak FVC values prior to first dose of randomized treatment. Peak FVC (0-3h) values were obtained within 0 - 3 hours after treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 19
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.268 (0.029) | 0.454 (0.028) | 0.474 (0.028) | 0.551 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.186, 95% CI [0.108 to 0.264], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.206, 95% CI [0.128 to 0.284], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.283, 95% CI [0.205 to 0.361], Standard Error of Mean 0.040 — Form 12 mcg minus Placebo

38. Secondary Outcome: Peak FVC (0-3h) Response After 6 Weeks
Description: as for outcome 37
Time Frame: as for outcome 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.202 (0.029) | 0.411 (0.028) | 0.433 (0.029) | 0.467 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.209, 95% CI [0.131 to 0.288], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.231, 95% CI [0.153 to 0.310], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.265, 95% CI [0.187 to 0.344], Standard Error of Mean 0.040 — Form 12 mcg minus Placebo

39. Secondary Outcome: Peak FVC (0-3h) Response After 12 Weeks
Description: as for outcome 37
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.194 (0.030) | 0.382 (0.029) | 0.432 (0.029) | 0.450 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.188, 95% CI [0.108 to 0.267], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.238, 95% CI [0.159 to 0.318], Standard Error of Mean 0.041 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.256, 95% CI [0.177 to 0.336], Standard Error of Mean 0.041 — Form 12 mcg minus Placebo

40. Secondary Outcome: Peak FVC (0-3h) Response After 24 Weeks
Description: as for outcome 37
Time Frame: as for outcome 22
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.207 (0.030) | 0.379 (0.029) | 0.414 (0.029) | 0.424 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.173, 95% CI [0.092 to 0.253], Standard Error of Mean 0.041 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.207, 95% CI [0.127 to 0.288], Standard Error of Mean 0.041 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.217, 95% CI [0.137 to 0.298], Standard Error of Mean 0.041 — Form 12 mcg minus Placebo

41. Secondary Outcome: Peak FVC (0-3h) Response After 48 Weeks
Description: as for outcome 37
Time Frame: as for outcome 23
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
Liter | 0.193 (0.031) | 0.344 (0.029) | 0.371 (0.030) | 0.416 (0.030)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.150, 95% CI [0.070 to 0.231], Standard Error of Mean 0.041 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.178, 95% CI [0.096 to 0.259], Standard Error of Mean 0.041 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.223, 95% CI [0.141 to 0.304], Standard Error of Mean 0.042 — Form 12 mcg minus Placebo

42. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) at Week 24
Description: Weekly mean pre-dose morning and evening PEFR. Results are from non-MMRM ANCOVA models by week, with Last observation carried forward (LOCF) up to each week. Fixed effects include treatment, tiotropium, strata and baseline.
Time Frame: Week 24
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 222 | 223 | 223
L/min
  morning PEFR (N=214, 212, 216, 218) | 196.429 (3.392) | 211.496 (3.420) | 211.428 (3.379) | 214.070 (3.373)
  evening PEFR (N=215, 211, 215, 221) | 202.256 (3.363) | 219.977 (3.408) | 220.727 (3.360) | 220.129 (3.332)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Comparison for Weekly mean morning PEFR; Test type: Superiority or Other; p = 0.0012, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 15.067, 95% CI 2-sided [5.962 to 24.173], Standard Error of Mean 4.639
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Comparison for Weekly mean morning PEFR; Test type: Superiority or Other; p = 0.0012, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 14.999, 95% CI [5.949 to 24.049], Standard Error of Mean 4.611
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Comparison for Weekly mean morning PEFR; Test type: Superiority or Other; p = 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 17.642, 95% CI 2-sided [8.610 to 26.673], Standard Error of Mean 4.601
Statistical Analysis 4: Comparison: Placebo vs Olo 5 mcg qd; Comparison for Weekly mean evening PEFR; Test type: Superiority or Other; p = 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 17.721, 95% CI 2-sided [8.680 to 26.762], Standard Error of Mean 4.606
Statistical Analysis 5: Comparison: Placebo vs Olo 10 mcg qd; Comparison for Weekly mean evening PEFR; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 18.471, 95% CI 2-sided [9.484 to 27.458], Standard Error of Mean 4.579
Statistical Analysis 6: Comparison: Placebo vs Form 12 mcg; Comparison for Weekly mean evening PEFR; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 17.873, 95% CI 2-sided [8.947 to 26.799], Standard Error of Mean 4.548

43. Secondary Outcome: Use of Rescue Medication at Week 24
Description: Mean number of puffs of rescue medication used per day (daytime/nighttime/total)
Time Frame: Week 24
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 217 | 212 | 216 | 221
Number of puffs
  Daytime | 1.364 (0.097) | 0.961 (0.099) | 1.037 (0.097) | 1.217 (0.097)
  Nighttime | 2.051 (0.125) | 1.449 (0.126) | 1.471 (0.125) | 1.701 (0.124)
  Total | 3.390 (0.196) | 2.399 (0.198) | 2.488 (0.196) | 2.917 (0.195)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Comparison for weekly mean daytime rescue use; Test type: Superiority or Other; p = 0.0026, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.403, 95% CI 2-sided [-0.665 to -0.141], Standard Error of Mean 0.133
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Comparison for weekly mean daytime rescue use; Test type: Superiority or Other; p = 0.0141, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.327, 95% CI 2-sided [-0.587 to -0.066], Standard Error of Mean 0.133
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Comparison for weekly mean daytime rescue use; Test type: Superiority or Other; p = 0.2677, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.147, 95% CI 2-sided [-0.406 to 0.113], Standard Error of Mean 0.132
Statistical Analysis 4: Comparison: Placebo vs Olo 5 mcg qd; Comparison for weekly mean nighttime rescue use; Test type: Superiority or Other; p = 0.0005, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.602, 95% CI 2-sided [-0.939 to -0.266], Standard Error of Mean 0.171
Statistical Analysis 5: Comparison: Placebo vs Olo 10 mcg qd; Comparison for weekly mean nighttime rescue use; Test type: Superiority or Other; p = 0.0007, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.580, 95% CI 2-sided [-0.914 to -0.247], Standard Error of Mean 0.170
Statistical Analysis 6: Comparison: Placebo vs Form 12 mcg; Comparison for weekly mean nighttime rescue use; Test type: Superiority or Other; p = 0.0391, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.350, 95% CI 2-sided [-0.683 to -0.018], Standard Error of Mean 0.169
Statistical Analysis 7: Comparison: Placebo vs Olo 5 mcg qd; Comparison for weekly mean daily (24h) rescue use; Test type: Superiority or Other; p = 0.0002, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.991, 95% CI 2-sided [-1.518 to -0.464], Standard Error of Mean 0.269
Statistical Analysis 8: Comparison: Placebo vs Olo 10 mcg qd; Comparison for weekly mean daily (24h) rescue use; Test type: Superiority or Other; p = 0.0008, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.902, 95% CI 2-sided [-1.426 to -0.378], Standard Error of Mean 0.267
Statistical Analysis 9: Comparison: Placebo vs Form 12 mcg; Comparison for weekly mean daily (24h) rescue use; Test type: Superiority or Other; p = 0.0758, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.473, 95% CI 2-sided [-0.994 to 0.049], Standard Error of Mean 0.266

44. Secondary Outcome: Patient's Global Rating (PGR) at 6 Weeks
Description: Patient's Global Rating (PGR) was a patient assessment of their health (respiratory condition) at each visit (compared to the day before they started study drug) and ranged from 1 (very much better) to 7 (very much worse).
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 194 | 216 | 212 | 206
score on a scale | 3.4 (0.1) | 3.0 (0.1) | 3.1 (0.1) | 3.1 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.4, 95% CI [-0.6 to -0.2], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0073, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0017, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Form 12 mcg minus Placebo

45. Secondary Outcome: Patient's Global Rating (PGR) at 12 Weeks
Description: as for outcome 44
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 194 | 216 | 212 | 206
score on a scale | 3.3 (0.1) | 3.0 (0.1) | 2.9 (0.1) | 3.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.4, 95% CI [-0.6 to -0.2], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0121, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Form 12 mcg minus Placebo

46. Secondary Outcome: Patient's Global Rating (PGR) at 24 Weeks
Description: as for outcome 44
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 194 | 216 | 212 | 206
score on a scale | 3.1 (0.1) | 2.9 (0.1) | 2.9 (0.1) | 3.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0320, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to -0.0], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0447, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to -0.0], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.1332, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to 0.0], Standard Error of Mean 0.1 — Form 12 mcg minus Placebo

47. Secondary Outcome: Patient's Global Rating (PGR) at 48 Weeks
Description: as for outcome 44
Time Frame: Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 194 | 216 | 212 | 206
score on a scale | 3.1 (0.1) | 3.0 (0.1) | 2.9 (0.1) | 2.9 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.4105, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.1, 95% CI [-0.3 to 0.1], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0584, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to 0.0], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.1006, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects, patient as random effect; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to 0.0], Standard Error of Mean 0.1 — Form 12 mcg minus Placebo

48. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 6 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 192 | 212 | 207 | 202
score on a scale | 0.995 (0.248) | 1.566 (0.236) | 1.660 (0.240) | 1.753 (0.243)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0882, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.571, 95% CI [-0.085 to 1.227], Standard Error of Mean 0.335 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0484, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.664, 95% CI [0.005 to 1.324], Standard Error of Mean 0.336 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.0252, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.758, 95% CI [0.094 to 1.421], Standard Error of Mean 0.338 — Form 12 mcg minus Placebo

49. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 12 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 192 | 212 | 207 | 202
score on a scale | 1.412 (0.252) | 1.792 (0.239) | 1.955 (0.242) | 1.805 (0.245)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2625, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.381, 95% CI [-0.285 to 1.047], Standard Error of Mean 0.340 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1109, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.543, 95% CI [-0.125 to 1.211], Standard Error of Mean 0.341 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.2507, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.394, 95% CI [-0.278 to 1.066], Standard Error of Mean 0.343 — Form 12 mcg minus Placebo

50. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 18 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 18
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 192 | 212 | 207 | 202
score on a scale | 1.665 (0.254) | 1.897 (0.240) | 2.099 (0.244) | 1.689 (0.246)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.4895, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.232, 95% CI [-0.439 to 0.902], Standard Error of Mean 0.342 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.2073, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.434, 95% CI [-0.240 to 1.107], Standard Error of Mean 0.344 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.9462, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.023, 95% CI [-0.653 to 0.700], Standard Error of Mean 0.345 — Form 12 mcg minus Placebo

51. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 32 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 32
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 192 | 212 | 207 | 202
score on a scale | 1.732 (0.257) | 1.898 (0.241) | 1.698 (0.247) | 1.966 (0.249)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.6309, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.166, 95% CI [-0.511 to 0.842], Standard Error of Mean 0.345 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.9227, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.034, 95% CI [-0.717 to 0.649], Standard Error of Mean 0.348 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.5030, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.234, 95% CI [-0.451 to 0.919], Standard Error of Mean 0.349 — Form 12 mcg minus Placebo

52. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 40 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 192 | 212 | 207 | 202
score on a scale | 1.952 (0.259) | 1.839 (0.241) | 1.887 (0.249) | 1.575 (0.251)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.7459, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.112, 95% CI [-0.793 to 0.568], Standard Error of Mean 0.347 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.8534, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.065, 95% CI [-0.753 to 0.623], Standard Error of Mean 0.351 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.5099, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.377, 95% CI [-1.068 to 0.314], Standard Error of Mean 0.352 — Form 12 mcg minus Placebo

53. Secondary Outcome: Mahler Transitional Dyspnea Index Focal Score at 48 Weeks
Description: as for outcome 3
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 192 | 212 | 207 | 202
score on a scale | 1.940 (0.259) | 2.035 (0.242) | 2.324 (0.250) | 2.047 (0.251)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.7850, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.095, 95% CI [-0.587 to 0.777], Standard Error of Mean 0.348 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.2755, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.383, 95% CI [-0.306 to 1.073], Standard Error of Mean 0.352 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.7618, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.107, 95% CI [-0.584 to 0.798], Standard Error of Mean 0.353 — Form 12 mcg minus Placebo

54. Secondary Outcome: Time to First Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (95% Confidence Interval); unit: Days
Groups:
- Placebo (Tiotropium): Matching Placebo delivered by the Respimat Inhaler - tiotropium use stratum
- Placebo (Non-tiotropium): Matching Placebo delivered by the Respimat Inhaler - non-tiotropium use stratum.
- Olo 5 mcg qd (Tiotropium): Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler - tiotropium stratum
- Olo 5 mcg qd (Non-tiotropium): Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler - non-tiotropium stratum
- Olo 10 mcg qd (Tiotropium): Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler - tiotropium stratum
- Olo 10 mcg qd(Non-tiotropium): Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler - non-tiotropium stratum
- Form 12 mcg (Tiotropium): Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler - tiotropium stratum
- Form 12 mcg (Non-tiotropium): Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler - non-tiotropium stratum
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium) | Form 12 mcg (Tiotropium) | Form 12 mcg (Non-tiotropium)
Number analyzed (Participants) | 57 | 168 | 60 | 167 | 58 | 167 | 58 | 169
Days | 143 [70.0 to 254.0] | 268 [149.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 136 [74.0 to 255.0] | 189 [115.0 to 262.0] | 134 [61.0 to 200.0] | 209 [109.0 to 290.0] | 223 [115.0 to 280.0] | 310 [207.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed.
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Olo 5 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.3424, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.162, 95% CI [0.843 to 1.603], Standard Error of Mean 0.190 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Non-tiotropium) vs Olo 10 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.3023, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.186, 95% CI [0.859 to 1.636], Standard Error of Mean 0.195 — Comparison of Olo 10 mcg qd to placebo across stratum
Statistical Analysis 3: Comparison: Placebo (Tiotropium) vs Form 12 mcg (Tiotropium); Test type: Superiority or Other; p = 0.3589, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.854, 95% CI [0.605 to 1.205], Standard Error of Mean 0.150 — Comparison of Form 12 mcg to placebo across stratum

55. Secondary Outcome: Time to First Chronic Obstructive Pulmonary Disease (CPOD) Exacerbation Leading to Hospitalization
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations required hospitalization. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium) | Form 12 mcg (Tiotropium) | Form 12 mcg (Non-tiotropium)
Number analyzed (Participants) | 57 | 168 | 60 | 167 | 58 | 167 | 58 | 169
Days | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed. | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed.
Statistical Analysis 1: Comparison: Placebo (Non-tiotropium) vs Olo 5 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.1910, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.818, 95% CI [0.734 to 4.503], Standard Error of Mean 0.841 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Non-tiotropium) vs Olo 10 mcg qd(Non-tiotropium); Test type: Superiority or Other; p = 0.2274, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.743, 95% CI [0.695 to 4.369], Standard Error of Mean 0.817 — Comparison of Olo 10 mcg qd to placebo across stratum
Statistical Analysis 3: Comparison: Placebo (Non-tiotropium) vs Form 12 mcg (Tiotropium); Test type: Superiority or Other; p = 0.5538, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.346, 95% CI [0.512 to 3.538], Standard Error of Mean 0.664 — Comparison of Form 12 mcg to placebo across stratum

56. Secondary Outcome: Time to First Moderate Chronic Obstructive Pulmonary Disease (CPOD) Exacerbation
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations did not lead to hospitalization but included treatment with antibiotics and/or systemic steroids. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium) | Form 12 mcg (Tiotropium) | Form 12 mcg (Non-tiotropium)
Number analyzed (Participants) | 57 | 168 | 60 | 167 | 58 | 167 | 58 | 169
Days | 150 [86.0 to 325.0] | 296 [215.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 239 [98.0 to 304.0] | 244 [154.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 175 [123.0 to 271.0] | 302 [213.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 280 [167.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed. | 270 [270.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed.
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Olo 5 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.5577, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.101, 95% CI [0.778 to 1.557], Standard Error of Mean 0.195 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Tiotropium) vs Olo 10 mcg qd (Tiotropium); Test type: Superiority or Other; p = 0.9423, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.017, 95% CI [0.714 to 1.448], Standard Error of Mean 0.184 — Comparison of Olo 10 mcg qd to placebo across stratum
Statistical Analysis 3: Comparison: Placebo (Tiotropium) vs Form 12 mcg (Tiotropium); Test type: Superiority or Other; p = 0.1097, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.735, 95% CI [0.502 to 1.076], Standard Error of Mean 0.143 — Comparison of Form 12 mcg to placebo across stratum

57. Secondary Outcome: Number of COPD Exacerbations
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria.
Time Frame: Baseline to end of study at week 48 visit
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: Number of COPD ex. per patient year
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 225 | 227 | 225 | 227
Number of COPD ex. per patient year | 0.5684 (0.0718) | 0.7117 (0.0793) | 0.6946 (0.0801) | 0.5098 (0.0649)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1729, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.2521, 95% CI [0.9060 to 1.7304], Standard Error of Mean 0.2064 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.2297, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.2220, 95% CI [0.8808 to 1.6954], Standard Error of Mean 0.2039 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.5354, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.8968, 95% CI [0.6353 to 1.2659], Standard Error of Mean 0.1575 — Form 12 mcg minus Placebo

58. Secondary Outcome: Number of COPD Exacerbations Requiring Hospitalization
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations required hospitalization.
Time Frame: Baseline to end of study at week 48 visit
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: Number of COPD ex. per patient year
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 225 | 227 | 225 | 227
Number of COPD ex. per patient year | 0.0554 (0.0249) | 0.1043 (0.0378) | 0.1324 (0.0493) | 0.0570 (0.0227)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2508, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.8821, 95% CI [0.6391 to 5.5430], Standard Error of Mean 1.0358 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1135, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 2.3877, 95% CI [0.8122 to 7.0194], Standard Error of Mean 1.3119 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.9611, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.0289, 95% CI [0.3268 to 3.2395], Standard Error of Mean 0.6013 — Form 12 mcg minus Placebo

59. Secondary Outcome: Number of Moderate Chronic Obstructive Pulmonary Disease (CPOD) Exacerbations
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations did not lead to hospitalization but included treatment with antibiotics and/or systemic steroids.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: Number of COPD ex. per patient year
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 225 | 227 | 225 | 227
Number of COPD ex. per patient year | 0.4765 (0.0645) | 0.5537 (0.0674) | 0.5114 (0.0654) | 0.3721 (0.0537)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.4002, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.1621, 95% CI [0.8187 to 1.6497], Standard Error of Mean 0.2075 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6983, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.0733, 95% CI [0.7503 to 1.5352], Standard Error of Mean 0.1957 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Test type: Superiority or Other; p = 0.2033, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 0.7810, 95% CI [0.5336 to 1.1433], Standard Error of Mean 0.1516 — Form 12 mcg minus Placebo

60. Secondary Outcome: Absolute Plasma Concentrations
Description: Absolute plasma concentrations of Olodaterol. Values presented are across visits and summarised into geometric means.
Time Frame: within 2 hours before first drug administration and 10 minutes post-dose at week 6, 12 and 18
Population: Pharmacokinetic set includes all patients in the treated set who had at least one valid olodaterol plasma concentration measurement after initial administration of study drug. This set is restricted to patients in either the Olodaterol 5 μg or 10 μg dose group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 0 | 178 | 205 | 0
pg/mL |  | 4.179 (60.300) | 7.246 (72.242) |

61. Secondary Outcome: Changes in Safety Parameters Related to Treatment
Description: Occurence of cardiac disorders and investigations related to treatment.
Time Frame: 48 weeks
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 225 | 227 | 225 | 227
percentage of participants
  Tachycardia | 0.4 | 0.0 | 0.0 | 0.9
  Arrhythmia | 0.0 | 0.4 | 0.0 | 0.0
  Atrial fibrillation | 0.4 | 0.0 | 0.0 | 0.4
  Atrioventricular block | 0.4 | 0.0 | 0.0 | 0.0
  Atrioventricular block first degree | 0.0 | 0.0 | 0.0 | 0.4
  Bundle branch block right | 0.0 | 0.4 | 0.0 | 0.0
  Palpitations | 0.4 | 0.0 | 0.0 | 0.4
  Ventricular extrasystoles | 0.4 | 0.0 | 0.0 | 0.0
  Electrocardiogram QT prolonged | 0.0 | 0.4 | 0.0 | 0.4
  Electrocardiogram T wave inversion | 0.0 | 0.0 | 0.0 | 0.4

62. Primary Outcome: Mahler Transitional Dyspnea Index Focal Score at 24 Weeks for Combined Analysis
Description: This outcome measure describes the combined analysis of the trials NCT00793624 and NCT00796653. Mahler Transitional Dyspnea Index (TDI) focal score measures 3 components of dyspnea that evoke dyspnea in daily living: Functional Impairment, Magnitude of Task, and Magnitude of Effort. The TDI measures the change from the baseline assessment ranging from -9 (most deterioration) to +9 (most improvement).
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg
Number analyzed (Participants) | 413 | 433 | 427 | 417
score on a scale | 1.471 (0.155) | 1.980 (0.175) | 1.996 (0.170) | 1.827 (0.168)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Olo 5mcg minus placebo; Test type: Superiority or Other; p = 0.0270, pattern mixture model; See Hogan, et. al. Hogan JW, Roy J, Korkontzelou C Tutorial in biostatistics:handling drop-out in longitudinal studies. Stat Med 23,1455-1497(2004); Mean Difference (Final Values) = 0.509, 95% CI [0.058 to 0.960], Standard Error of Mean 0.230 — Based on a pattern mixture model with four patterns based on time of dropout (i.e., day of last observed data) 1) day 43 or day 85, 2) day 127 or day 169, 3) day 225 or day 281, 4) day 337
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Olo 10 mcg minus placebo; Test type: Superiority or Other; p = 0.0203, pattern mixture model — See Hogan, et. al. Hogan JW, Roy J, Korkontzelou C Tutorial in biostatistics:handling drop-out in longitudinal studies. Stat Med 23,1455-1497(2004); Mean Difference (Final Values) = 0.525, 95% CI [0.082 to 0.967], Standard Error of Mean 0.226 — [estimate comment as in outcome 62, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg; Form 12mcg minus placebo; Test type: Superiority or Other; p = 0.1166, pattern mixture model; [statistical method as in outcome 62, analysis 1]; Mean Difference (Final Values) = 0.355, 95% CI [-0.088 to 0.799], Standard Error of Mean 0.226 — [estimate comment as in outcome 62, analysis 1]

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Placebo | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd | Form 12 mcg
Serious Adverse Events (participants affected / at risk) | 31/225 | 33/227 | 26/225 | 33/227
Other Adverse Events (participants affected / at risk) | 83/225 | 100/227 | 96/225 | 83/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=225) | Olodaterol (Olo) 5 mcg qd (N=227) | Olodaterol (Olo) 10 mcg qd (N=225) | Form 12 mcg (N=227)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 3 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0 | 0
Ophthalmoplegia (Eye disorders) | 0 | 0 | 0 | 1
Parophthalmia (Eye disorders) | 1 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatic insufficiency (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Hernia (General disorders) | 0 | 1 | 0 | 0
Mass (General disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 0 | 1 | 1
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 6 | 8 | 3
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound abscess (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 13 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dental care (Surgical and medical procedures) | 0 | 1 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=225) | Olodaterol (Olo) 5 mcg qd (N=227) | Olodaterol (Olo) 10 mcg qd (N=225) | Form 12 mcg (N=227)
Nasopharyngitis (Infections and infestations) | 15 | 22 | 25 | 23
Upper respiratory tract infection (Infections and infestations) | 15 | 17 | 11 | 11
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 51 | 67 | 62 | 53
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 13 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 13 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication